CLINICAL TRIAL: NCT07339150
Title: MiREA, a mHealth Intervention to Reduce Health Disparities by Improving Access to Mandated College Students With Problematic Alcohol and Marijuana Use
Brief Title: MiREA-AC for Reducing Problematic Alcohol and Marijuana Use in College Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: mHealth Systems Inc. (Industry)
Collaborators: Boston Children's Hospital (Other); University of North Carolina, Charlotte (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MiREA-AC STTR Phase I; R41MD019586 (NIH)
Record Dates: First submitted 2025-09-29; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Alcohol Misuse; Cannabis Misuse
Keywords: mHealth; smart phone application; alcohol misuse; Cannabis misuse; health-seeking behaviors
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental arm which received the intervention (Experimental): experimental arm receives two week dose of the MiREA intervention
  Interventions: Behavioral: Motivational Intervention Reduction through Ecological Application (MiREA-A). MiREA-AC-- the expanded MiREA-A,

INTERVENTIONS:
Behavioral: Motivational Intervention Reduction through Ecological Application (MiREA-A). MiREA-AC-- the expanded MiREA-A, — MiREA-A, is based on Brief Motivational Interventions (BMI) core concepts to bring change in Alcohol & Cannabis use. It examines why someone uses substances and provides personalized feedback on consumption and consequences, social norms, and challenges. Feedback is designed to reveal discrepancies between students' use and goals.

SUMMARY:
The goal of this STTR Phase I funded study is to address the urgent need for an effective primary prevention approach to the problem of heavy episodic drinking and cannabis misuse among mandated college students. Smartphone app interventions are expanding and can offer accessible, scalable, and cost-effective tools. The study will be used to attune a successful evidence-based mHealth smartphone (SP) application (MiREA-AC) focused on alcohol and Cannabis misuse by college students with enhanced content to promote health-seeking behaviors. To test and disseminate the adapted prototype (MiREA-AC), a multisite pilot trial will be conducted to obtain data on the intervention's usability and feasibility in modifying alcohol and cannabis use.

DETAILED DESCRIPTION:
MiREA-A intervention is effective with alcohol. MiREA-AC-- the expanded MiREA-A -- has three new features: (1) cannabis content, (2) enhanced UX/UI interface, and (3) information modules for administrative reporting obligations. The study has two aims, as detailed in the following sections - a pilot trial for feasibility and customer discovery for features refinement, commercialization dissemination, reach, and sustainability.

Aim 1: Determine usability, feasibility, and preliminary efficacy of the MiREA-AC intervention (months 1-12); the study will: a) conduct alpha theater and field testing (months 1-3, n=10) at two U.S. campuses to ensure acceptability of the app's three new features; b) conduct a multi-site pilot feasibility trial (months 3-12, n=50) at six U.S. campuses. Metric 1: MiREA-AC refinement completed. Preliminary pilot feasibility testing was conducted on six U.S. campuses (month 12).

MiREA -AC app is designed to be delivered over two weeks, consistent with the delivery of a two-session in-person BMI. The features are delivered in modules which are activated when they are downloaded to the participants' smartphones. Users can then navigate the nine modules of the app with user-friendly directions. The MiREA app has been expanded to include integrated alcohol and cannabis features (MiREA-AC). The eight integrated features are Intro Video, Daily Log, Virtual Coach, Text Messages, Personalized Feedback, Gaming (Learn More), My Strategies, and Where to Go. Theoretical Framework: MiREA-AC incorporates three main theoretical approaches to reduce alcohol and Cannabis misuse in young adults. EMIs can combine ecological momentary assessment (EMA) with real-time delivery to facilitate change. Motivational Interviewing (used in BMIs) is a conversational approach that guides ambivalent clients toward change. According to the Transtheoretical Model (TTM), a leading theory of health behavior change, there are five stages of change: precontemplation, contemplation, preparation, action, and maintenance. As in the study team's prior work, the IDEAS framework was used to guide MiREA-AC development.

Alpha Testing: Theater testing and field-testing during development (months 1-3) will examine the accuracy and address potential technical issues of the developed app. Ten mandated students will be recruited at two U.S. campuses (UNC Charlotte and USC). After an initial in-person session that orients the student to the study, facilitators will demonstrate and explain the app's features (e.g., coach, personalized feedback, alcohol/cannabis tracking) to participants. Participants will use MiREA-AC for two weeks and then complete brief surveys for their reactions to the smartphone app. The APP usage data will be collected, including how often and how much time each app component is used and any mistakes or errors appearing during their use. The study team will correct the errors and make necessary changes to the app based on students' feedback on the ease of use, helpfulness, and overall satisfaction. Pilot Study Sites: A pilot study will then be implemented to assess feasibility and accessibility (months 3-12). Pilot sites will consist of six public and private colleges with diverse backgrounds. All participate in the National Collegiate Health Association survey, which indicates the frequency of drinking and heavy drinking at their schools are consistent with national findings. The target is to enroll 50 eligible students and retain at least 75% at two weeks.

Pilot Study Eligibility: Inclusion criteria: 18- to 25-year-old college students mandated to programming for alcohol and drug policy violations. Positive screening for alcohol use in the past 90 days. A score ≥ 4 on the Alcohol Use Disorders Identification Test-Alcohol Consumption Questions (AUDIT-C), the recommended maximum for drinking among mandated college students.

Pilot Trial Study Design: After enrollment, facilitators (site logistics managers) will build rapport with participants, have them download the MiREA-AC app to their phones, and teach them how to use the app and other APP features. The students will be instructed to use the app for two weeks, during which the participants will receive constant personalized feedback. It is hypothesized that mHealth Systems' real-time "push" technologies will raise students' consciousness and reinforce substance use behavior change.

MiREA-AC Baseline. Eligible students enrolled in the study will use the app to complete baseline questionnaires regarding their substance use history, its consequences, and their demographic characteristics. During the two-week treatment period, APP usage data will be collected, including how often and how much time each module is used and the number of personalized messages sent to them.

Two-Week Visit: Participants will give feedback on the app's usability and acceptability as well as issues related to their alcohol and cannabis use and consequences. Six-Week Follow-up: Participants will be followed up and asked to report the student's alcohol and cannabis use and consequences.

Measures. Primary endpoints for assessing the feasibility of the app include participating rate (the number of enrolled participants/the number of eligible students asked to participate), retention rate (proportion of participants who complete two-week visit), treatment adherence (the frequency and length of each module of the app being used during the treatment). Satisfaction measures include outcomes from a satisfactory survey and the Usefulness, Satisfaction, and Ease of Use questionnaire at the end of the two-week treatment.56 Statistical Plan and Data Analysis: The participation and retention rates will be reported at two weeks and include summary statistics of the intervention adherence data since there is little existing knowledge of the feasibility of mHealth intervention for cannabis use and, therefore no existing golden standard for feasibility. With feedback responses to the satisfactory and USE questionnaire, the potential efficacy of the APP will be explored by comparing the participant's substance usage and consequences between baseline and follow-up.

Aim 2: Examine key customer needs by engaging with a Stakeholders Advisory Board (SAB, n=50, months 1-12) composed of health wellness staff, administrators, and minority representatives from HBCUs and ARC socioeconomically disadvantaged colleges and universities and engage the SAB in the integration of MiREA-AC prototype within their mandated programs. Metric 2: SAB meetings completed (by month 12) with representatives (N=50) from six diverse campuses; summary report of customer needs.

ELIGIBILITY:
Inclusion Criteria:

* College student, alcohol consumption in past 90 days

Exclusion Criteria:

* non-college student, no alcohol use in the past 90 days

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Eligible participants solicited | 6 Months
  Number of eligible participants of the study that we reach out to.
Enrolled | 6 months
  Number of eligible participants enrolled
2-week intervention | 6 months
  Number of enrolled participants who complete the 2-week intervention.
Usability score | 6 months
  Usability score by a mHealth App Usability Questionnaire (MAUQ)56 at 2-week.The USE 26-item questionnaire is widely used for measuring usefulness and ease of use. Each factor is designed to measure the user satisfaction and ease of learning. It was designed as a 7-point Likert scale questionnaire, where 1 = strongly disagree and 7 = strongly agree. Usability is measured on three dimensions: Usefulness (4 items), Satisfaction (7 items), and Ease of use (15 items). Sample questions include, "I am satisfied with it", "it is useful", "it meets my needs" "it is a pleasure to use "and "I learned to use it quickly.
Satisfactory Survey | 6 months
  Outcomes of a team-designed satisfactory survey at 2 weeks.

SECONDARY OUTCOMES:
Daily alcohol use | 6 months
  Daily alcohol use by Modified Daily Drinking Questionnaire (DDQ),55 during the intervention.DDQ is a 7-item face-valid instrument measuring alcohol consumption. It assesses alcohol patterns, including quantity, frequency of use, and peak drinking events, on a daily basis over a typical week; these are then averaged over the past month. DDQ has been modified to collect descriptive demographic information, including gender, race/ethnicity, and age. The mean number of drinks per week is calculated by multiplying the amount by the frequency of drinking. The DDQ has been validated for use with college students.
Alcohol disorders identification | 6 months
  Alcohol Use Disorders Identification Test (AUDIT-C)52,53,54 at baseline, 2-week, and 6-week.Description: AUDIT is a three-question screen used to identify alcohol misuse. It is scored on a scale of 0-12 points (scores of 0 reflect no alcohol use in the past year). The AUDIT-C has performed better than the AUDIT and CAGE screen in identifying heavy drinkers who might benefit from brief interventions56 and it has been validated among college students as a screening tool.49,50 An AUDIT-C cutoff score of 4 or greater demonstrated a sensitivity of 92.6% and a specificity of 86.3% in detecting risky drinkers among college students.
Alcohol consequences | 6 months
  Alcohol consequences will be assessed by the B-YAACQ at baseline, 2-week, and 6-week.The B-YAACQ will be used to assess the results of the past month's alcohol consequences at each time point. This is a 24-question screen used to identify alcohol consequences. Outcome scores range from 0 to 24. The 30-day B-YAACQ has demonstrated high internal consistency (alpha=.89) for evaluating changes in alcohol consequences.
Alcohol Consequence Questionnaire | 6 months
  Brief Young Adult Alcohol Consequence Questionnaire (B-YAACQ) at baseline, 2-week, and 6-week.
Readiness Ruler | 6 weeks
  Readiness Ruler: a scale with a 0-to-10 range, with a minimum value of 0 and a maximum value of 10, to help people evaluate the importance of changing substance use behaviors. It helps individuals and service providers gauge where someone is on a spectrum from worse "0" "not prepared to change" to better "10" "already changing" by using two simple questions with a scale of 0 to 10 for importance and confidence.
Comprehensive effects of Alcohol | 6 months
  Brief Comprehensive Effects of Alcohol Scale at baseline, 2-week, and 6-week.The BCEAS is a 15-item measure that assesses positive (e.g., "I would act sociable") and negative (e.g., "I would feel dizzy") alcohol expectancies (i.e., expectations about the effects of alcohol use) and valuations of these expectancies (the extent to which a student believes a certain effect to be 'good' or 'bad'). Students report their level of agreement with each expectancy statement using a 4-point scale (1 = Disagree to 4 = Agree), and their valuations of these expectancy outcomes using a 5-point scale (1 = Bad to 5 = Good).
Marijuana consequences | 6 months
  Marijuana consequences will be assessed by the Marijuana Problems Scale (MPS) at baseline, 2-week, and 6-week.: Marijuana Problems Scale (MPS) is a 19-item measure of the number and severity of marijuana problems during the past 90 days. Domains include psychological, social, occupational, and legal consequences with response options on a 3-point scale (no problem, minor problem, serious problem).
Marijuana effect expectancies | 6 months
  Marijuana Effect Expectancies Questionnaire (MEEQ), at baseline, 2-week, and 6-week.A 48-item questionnaire (5-pt Likert scale) assesses beliefs about possible consequences of marijuana with six scales. We will test negative outcomes expectancies: global negative effects (GN) and cognitive/behavioral impairment (CBI), as well as relaxation/tension reduction expectancies (TR), as moderators of the relationship between negative affect and marijuana use/problems/dependence.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of North Carolina, Charlotte, Charlotte, North Carolina
  - University of South Carolina, Columbia, South Carolina

IPD SHARING:
Plan to Share IPD: Undecided
Sharing plans are not yet determined.